CLINICAL TRIAL: NCT03352258
Title: Effect of Low Dose Radiotherapy on Brain Amyloidosis in the Treatment of Alzheimer's Disease: a Randomized Pilot Study
Brief Title: Effect of Low Dose Radiotherapy on Brain Amyloidosis in the Treatment of Alzheimer's Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Valentina Garibotto (Other)
Responsible Party: Sponsor-Investigator, Valentina Garibotto, Pr, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-01715
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; Amyloid; Radiotherapy
MeSH Terms: conditions — Alzheimer Disease | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: Randomized, monocentric, prospective pilot study, pre- and post-intervention intraindividual comparison in the treated arm comparison of changes in neuropsychological performance in the treated and observational arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observation (No Intervention): Subjects in this arm will only be followed and not treated (observational arm)
- Treatment arm (Experimental): Subjects will receive a low dose brain radiotherapy
  Interventions: Radiation: Low dose radiotherapy

INTERVENTIONS:
Radiation: Low dose radiotherapy — 10 Gy in 5 fractions of 2 Gy on 5 consecutive days
  Arms: Treatment arm

SUMMARY:
Alzheimer's Disease (AD) is the most frequent neurodegenerative disease associated with dementia, with a constantly increasing prevalence associated with an aging population. Amyloid deposition is considered the first molecular event occurring in AD: as already showed in an animal model, a low-dose radiotherapy (RT) course is capable of reducing AD-associated amyloid-β plaques and improve cognitive function. This pilot study wishes to investigate in 10 patients with a diagnosis of prodromal or early probable AD and with evidence of amyloid pathology the effectiveness of a short course low dose RT radiotherapy to reduce amyloid deposits in the human brain using molecular imaging (18F-Florbetapir) to show the effectiveness of the treatment on the specific target.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the clinical trial and give an informed consent
* Clinical diagnosis of prodromal AD, or mild or moderate AD
* Ability to undergo neurocognitive assessment at baseline visit, alone or accompanied by a caregiver
* Amyloid PET scan positivity
* Ability to follow the 5-days RT regiment, alone or accompanied by a caregiver

Exclusion Criteria:

* Inclusion in another disease modifying clinical trial
* Previous therapeutic brain irradiation
* Evidence of vascular cognitive impairment on Magnetic Resonance Imaging (MRI) (Fazekas score >1 and Wahlund score >=10/30)
* Oncologic disease (excluding skin cancer) active or in remission from less than 5 years
* Evidence of substance abuse (alcohol and/or other drugs) with a dependence during the previous 12 months (DSM-IV criteria)
* Presence of subdural hygroma's, subdural hematomas or hydrocephalus
* Significant psychiatric comorbidity as assessed during the clinical evaluation by the neurologist/geriatrician in charge
* Active or recent (within 3 months) cerebral infection/haemorrhage
* Immunocompromised status
* Prior history of seizure
* Dermatological skin disease of the scalp
* Women who are pregnant or breast feeding or who intend to become pregnant during the course of the study;
* Lack of safe contraception, defined as: female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse event associated with low dose brain RT | 12 months from end of RT
  Assess the number of patients who report adverse events
Change in brain amyloid deposits | 8-12 weeks from end of RT
  Assess intra-individual change in a quantitative measure of amyloid deposits on PET imaging (Standard Uptake Value ratio) SUVR between amyloid PET scans before and after low dose brain RT

SECONDARY OUTCOMES:
Neuropsychological performances | 6 months after inclusion
  Neurocognitive tests (assessing verbal and non-verbal memory, attention, executive function, praxis function, visuospatial functions, and language) to evaluate changes after low dose RT, as compared with a population of 10 subjects followed up clinically

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Garibotto, Pr, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided